CLINICAL TRIAL: NCT06085144
Title: Prospective Evaluation of Emgality (Galcanezumab) in Breastmilk in Adult Women With Migraine
Brief Title: Emgality for Migraine in Breastmilk
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: Emgality in breast milk
Record Dates: First submitted 2023-10-04; First posted 2023-10-16 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Migraine
Keywords: Emgality; Galcanezumab; Migraine; Breastmilk; Milk; Breastfeeding; Pregnancy; Postpartum; Monoclonal Antibodies
MeSH Terms: conditions — Migraine Disorders; Breast Feeding | interventions — galcanezumab; erenumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Participants will pump and provide up to 8 breastmilk samples (15mL volume each), at specific timepoints over up to 2 treatment cycles (before treatment 1; 24hours, 7d, 28d post treatment 1; 24hours, 7d, 28d post treatment 2 and 7d post treatment 3). Samples will be shipped in an insulated container with gel packs to maintain temperature via FedEx priority overnight shipping to our Laboratory at UCSF and stored in a -80 °C degrees freezer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Galcanezumab: Postpartum women both nursing and receiving treatment for migraine with galcanezumab.
  Interventions: Drug: Galcanezumab

INTERVENTIONS:
Drug: Galcanezumab — Receiving either 120mg or 300mg injections.
  Other Names: Emgality

SUMMARY:
The goal of this project is to evaluate galcanezumab transfer into maternal breastmilk, and to evaluate infant (growth, development, constipation, colic, infections) and maternal (headache) outcomes for dyads in which the mother was treated with galcanezumab and to compare outcomes for infants who were or were not breastfed after maternal treatment.

In this prospective observational study, the study team proposes to prospectively collect serial milk samples from 30 adult women who are treated with galcanezumab for migraine. Mothers who are interested in participating will be connected with us, the main clinical site, by neurologists across the USA. Mothers must carry a diagnosis of migraine, be aged 18-45 years, and be between 14 days and 9 months postpartum, and still nursing, at the time of enrollment.

This study will fill a significant unmet need as women of childbearing potential are over-represented in the migraine population, and yet they are excluded from clinical trials of migraine treatments during pregnancy and lactation.

DETAILED DESCRIPTION:
Galcanezumab will be prescribed clinically by the treating clinician, i.e., no drug will be provided by the study. This treatment may be prescribed in several clinical scenarios:

* Patient with established migraine history, treated with galcanezumab prior to pregnancy, who plans to resume the medication post partum
* Patient with established migraine history, who experiences migraines postpartum and who has previously been "failed by", or intolerant to, other first-line prophylactic medications
* Patient with established migraine history, who warrants said treatment trial otherwise, at the discretion of the prescribing clinician

Interested participants will be contacted by our UCSF coordinator, sign an informed consent form, and receive instructions for milk collection. A pamphlet on effective birth control will be provided to all enrollees (https://owh-wh-d9-dev.s3.amazonaws.com/s3fs-public/documents/fact-sheet-birth-control-methods.pdf), as well as OCT-available at-home pregnancy tests.

Mothers will complete questionnaires relating to their infants, at 6M and 12M postpartum (Ages and Stages, colic, etc.) and will sign a release form for us to obtain and review infant health records up to 12 months post-delivery to calculate: growth, infections, incidence of constipation or infant colic.

Milk collection:

Participants will pump and provide up to 8 samples (15mL volume each), at specific timepoints over up to 2 treatment cycles (before treatment 1; 24hours, 7d, 28d post treatment 1; 24hours, 7d, 28d post treatment 2 and 7d post treatment 3). Samples will be shipped in an insulated container with gel packs to maintain temperature via FedEx priority overnight shipping to our Laboratory at UCSF and stored in a -80 °C degrees freezer.

Sample assays:

Samples will be batch analyzed using enzyme immunoassay at (1) interim report after 15 sets received and (2) final report after all 30 sets received. The study team has worked with MarinBio who are experts in measuring biologics.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Childbearing age (18-45)
* Established diagnosis of migraine
* Status post uncomplicated delivery (no long-term maternal complications)
* No prolonged (>3 night) NICU stay for infant
* Between 14 days and 9 months postpartum, and still nursing, at the time of enrollment
* Planning to receive galcanezumab postpartum
* Suitable candidate to receive galcanezumab postpartum, at discretion of prescribing clinician

Exclusion Criteria:

* Contraindications to breastfeeding, such as prior surgery or infant contraindications
* Contraindications to galcanezumab or insurance coverage
* Use of gepants
* Moderately Severe or Severe Depression as established by the PHQ9 screen (i.e. score 15 or above)
* Pregnant or planning pregnancy in the coming 6M
* Patients with severe mastitis will not be enrolled; should mastitis occur during the study, this will be included as a covariate and results analyzed accordingly
* Patients of infants with severe medical issues identified in the health record (developmental issues, delivery issues, concomitant medications)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Mothers must carry a diagnosis of migraine, be aged 18-45 years, and be between 14 days and 9 months postpartum, and still nursing, at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Determine emgality concentration in mature breastmilk | 12 months
  Levels of galcanezumab (μg/mL) in the breastmilk of women at the selected timepoints before and after each treatment (24H pre, 24H post, 7D post, 28D post). For the third treatment, only 7D post will be collected. This outcome will be measured by breastmilk concentration (μg/mL).
Determine average emgality concentration in mature breastmilk | 12 months
  Levels of galcanezumab (μg/mL) in the breastmilk of women at the selected timepoints before and after each treatment (24H pre, 24H post, 7D post, 28D post). For the third treatment, only 7D post will be collected. This outcome will be measured by average breastmilk concentration (CAVE, determined using pharmacokinetic methods).
Determine maximum emgality concentration in mature breastmilk | 12 months
  Levels of galcanezumab (μg/mL) in the breastmilk of women at the selected timepoints before and after each treatment (24H pre, 24H post, 7D post, 28D post). For the third treatment, only 7D post will be collected. This outcome will be measured by maximum concentration of galcanezumab in breastmilk (CMAX).
Determine average emgality dose to infants through mature breastmilk in a 24-hour period | 12 months
  Levels of galcanezumab (μg/mL) in the breastmilk of women at the selected timepoints before and after each treatment (24H pre, 24H post, 7D post, 28D post). For the third treatment, only 7D post will be collected. This outcome will be measured by absolute average galcanezumab dose to the infant in a 24-hour period.
Determine maximum emgality dose to infants through mature breastmilk in a 24-hour period | 12 months
  Levels of galcanezumab (μg/mL) in the breastmilk of women at the selected timepoints before and after each treatment (24H pre, 24H post, 7D post, 28D post). For the third treatment, only 7D post will be collected. This outcome will be measured by maximum galcanezumab dose to the infant in a 24-hour period.
Determine average relative infant dose of emgality in mature breastmilk | 12 months
  Levels of galcanezumab (μg/mL) in the breastmilk of women at the selected timepoints before and after each treatment (24H pre, 24H post, 7D post, 28D post). For the third treatment, only 7D post will be collected. This outcome will be measured by average relative infant dose (RIDAVE).
  The investigators hypothesize that given that galcanezumab is an IgG mAb, it will similarly show very low concentrations, and acceptable relative infant dose (RID) (<1%).
Determine maximum relative infant dose of emgality in mature breastmilk | 12 months
  Levels of galcanezumab (μg/mL) in the breastmilk of women at the selected timepoints before and after each treatment (24H pre, 24H post, 7D post, 28D post). For the third treatment, only 7D post will be collected. This outcome will be measured by maximum relative infant dose (RIDMAX).
  The investigators hypothesize that given that galcanezumab is an IgG mAb, it will similarly show very low concentrations, and acceptable relative infant dose (RID) (<1%).

SECONDARY OUTCOMES:
Obtain information on newborn developmental milestones at 6 months of life | 6 months
  The Ages and Stages Questionnaire, third edition, (ASQ-3) will be completed by participating mothers at the following timepoints postpartum, to determine the developmental age of infants at 6 months. The questionnaire scores 5 areas of development: Communication, Gross Motor, Fine Motor, Problem Solving and Personal-Social. Cumulative scores range from 0 to 60. Higher scores indicate more positive outcomes. Each version of the ASQ-3 has different cutoff scores that indicate whether the child's development appears to be on schedule, requires monitoring or requires further assessment. (Above and Monitoring Ranges indicate on schedule infant development for age).
Obtain information on newborn developmental milestones at 12 months of life | 12 months
  The Ages and Stages Questionnaire, third edition, (ASQ-3) will be completed by participating mothers at the following timepoints postpartum, to determine the developmental age of infants at 12 months. The questionnaire scores 5 areas of development: Communication, Gross Motor, Fine Motor, Problem Solving and Personal-Social. Cumulative scores range from 0 to 60. Higher scores indicate more positive outcomes. Each version of the ASQ-3 has different cutoff scores that indicate whether the child's development appears to be on schedule, requires monitoring or requires further assessment. (Above and Monitoring Ranges indicate on schedule infant development for age).
Obtain information on newborn adjusted length until 12 months of life | 12 months
  Newborn adjusted length (in cm) will be collected by manual review of infant medical records at all visits occurring in the first 12 months of life.
Obtain information on newborn weight until 12 months of life | 12 months
  Newborn weight (in kg) will be collected by manual review of infant medical records at all visits occurring in the first 12 months of life.
Obtain information on newborn head circumference until 12 months of life | 12 months
  Newborn head circumference (in cm) will be collected by manual review of infant medical records at all visits occurring in the first 12 months of life.
Obtain information on the number of newborn infections until 12 months of life | 12 months
  The number of and nature of each newborn infections will be collected by manual review of infant medical records at all visits occurring in the first 12 months of life.
Obtain information on number of instances of newborn constipation including medications or interventions until 12 months of life | 12 months
  The number of instances of newborn constipation along with any relevant evidence will be collected by manual review of infant medical records at all visits occurring in the first 12 months of life.
Determine time to peak levels of galcanezumab in breastmilk | 12 months
  Levels of galcanezumab (μg/mL) in the breastmilk of women at the selected timepoints before and after each treatment (24H pre, 24H post, 7D post, 28D post). For the third treatment, only 7D post will be collected. The average peak level of galcanezumab concentration will be determined from this.
Determine headache severity surrounding the participants' galcanezumab treatments | 12 months
  The maternal migraine diary will be completed by participating mothers in the months surrounding their galcanezumab treatments. It tracks headache severity by asking participants to self-report their percieved headache severity on a scale of 0-10 daily.
Determine the number of days with headaches surrounding the participants' galcanezumab treatments | 12 months
  The maternal migraine diary will be completed by participating mothers in the months surrounding their galcanezumab treatments. It tracks headache dats by asking participants to self-report whether or not they experienced at least one migraine daily.
Determine what acute migraine medications were used by participants surrounding their galcanezumab treatments | 12 months
  The maternal migraine diary will be completed by participating mothers in the months surrounding their galcanezumab treatments. It tracks acute medication use by asking participants to self-report what acute medications they use to manage their migraines and when.

CONTACTS AND LOCATIONS:
Overall Officials: Riley Bove, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LaHue SC, Gelfand AA, Bove RM. Navigating monoclonal antibody use in breastfeeding women: Do no harm or do little good? Neurology. 2019 Oct 8;93(15):668-672. doi: 10.1212/WNL.0000000000008213. Epub 2019 Sep 6. PMID 31492717
- [Background] Krysko KM, LaHue SC, Anderson A, Rutatangwa A, Rowles W, Schubert RD, Marcus J, Riley CS, Bevan C, Hale TW, Bove R. Minimal breast milk transfer of rituximab, a monoclonal antibody used in neurological conditions. Neurol Neuroimmunol Neuroinflamm. 2019 Nov 12;7(1):e637. doi: 10.1212/NXI.0000000000000637. Print 2020 Jan. PMID 31719115
- [Background] Proschmann U, Haase R, Inojosa H, Akgun K, Ziemssen T. Drug and Neurofilament Levels in Serum and Breastmilk of Women With Multiple Sclerosis Exposed to Natalizumab During Pregnancy and Lactation. Front Immunol. 2021 Aug 26;12:715195. doi: 10.3389/fimmu.2021.715195. eCollection 2021. PMID 34512637